CLINICAL TRIAL: NCT03990181
Title: Testing the Efficacy of a Natural Polyphenol Supplement to Inhibit Dietary Iron Absorption in Subjects With Hereditary Hemochromatosis: a Stable Isotope Study
Brief Title: Inhibiting Dietary Iron Absorption in Subjects With Hereditary Hemochromatosis by a Natural Polyphenol Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Instituto de Investigação em Imunologia (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Head of the Laboratory of Human Nutrition, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FePPHH
Record Dates: First submitted 2019-06-09; First posted 2019-06-18 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Iron Metabolism Disorders; Iron Overload; Polyphenols
MeSH Terms: conditions — Iron Metabolism Disorders; Iron Overload | interventions — N-(3-pyridyl)-3-phenylsuccinimide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meal & natural polyphenol supplement (NPPS) (Experimental): A meal, labelled with stable iron isotope as ferrous sulphate, consumed with the natural polyphenol supplement
  Interventions: Dietary Supplement: meal matrix & NPPS
- Drink & natural polyphenol supplement (Experimental): A drink, labelled with stable iron isotope as ferrous sulphate, consumed with the natural polyphenol supplement
  Interventions: Dietary Supplement: no-matrix & NPPS
- Meal & control supplement (CS) (Placebo Comparator): A meal, labelled with stable iron isotope as ferrous sulphate, consumed with a control supplement
  Interventions: Dietary Supplement: meal matrix & CS
- Drink & control supplement (Placebo Comparator): A drink, labelled with stable iron isotope as ferrous sulphate, consumed with a control supplement
  Interventions: Dietary Supplement: no-matrix & CS

INTERVENTIONS:
Dietary Supplement: meal matrix & NPPS — Test meal consumed with the natural polyphenol supplement
  Arms: Meal & natural polyphenol supplement (NPPS)
Dietary Supplement: meal matrix & CS — Test meal consumed with the control supplement
  Arms: Meal & control supplement (CS)
Dietary Supplement: no-matrix & NPPS — Test drink consumed with the natural polyphenol supplement
  Arms: Drink & natural polyphenol supplement
Dietary Supplement: no-matrix & CS — Test drink consumed with the control supplement
  Arms: Drink & control supplement

SUMMARY:
Polyphenolic compounds are very strong Inhibitors of non-heme iron absorption, as they form insoluble complexes with ferrous iron. Patients with hereditary hemochromatosis (HH) have an increased intestinal non-heme iron absorption due to a genetic mutation in the regulatory pathway, leading to excess iron in the body. This study investigates the inhibitory effect of a natural polyphenol Supplement in participants with HH.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for C282Y mutation in HFE (hemochromatosis) gene
* Written informed consent
* Age 18-65 y
* Not pregnant or lactating
* Body weight < 75 kg
* Body mass index (BMI) between 18.5 and 25 kg/m2
* No acute illness/infection (self-reported)
* No metabolic or gastrointestinal disorders, eating disorders or food allergy to the ingredients of the test meal (self-reported)
* No scheduled phlebotomy throughout the study period
* The last phlebotomy will be at least 4 weeks prior first test meal administration
* No use of medications affecting iron absorption or metabolism during the study
* No intake of mineral/vitamin supplements 2 weeks before the first study day and during the study
* Participation in any other clinical study within the last 30 days
* Expected to comply with study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after administration of a test meal/drink including iron isotopes
change from baseline in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after administration of a test meal/drink including iron isotopes

SECONDARY OUTCOMES:
Serum Ferritin concentration (µg/L) | baseline, weeks 2, and 4
  to assess iron status
Serum iron concentration (µg/dL) | baseline, weeks 2, and 4
  to assess iron status
Soluble transferrin receptor (mg/L) | baseline, weeks 2, and 4
  to assess iron status
Transferrin saturation in % | baseline, weeks 2, and 4
  to calculate percent of transferrin that has iron bound to it; Plasma iron and transferrin saturation will be combined to calculate transferrin saturation (ratio)
Hemoglobin (g/dL) | baseline, weeks 2, and 4
  to assess blood volume based on weight, height, and Hb.
C-reactive Protein (mg/L) | baseline, weeks 2, and 4
  identify acute inflammation
alpha-1-glycoprotein (g/L) | baseline, weeks 2, and 4
  identify chronic inflammation
Serum Hepcidin (nM) | baseline, and weeks 2
  the major regulator of non-heme iron absorption

CONTACTS AND LOCATIONS:
Locations (2):
- Porto University Hospital Center, Porto, Portugal
- Laboratory of Human Nutrition ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buerkli S, Salvioni L, Koller N, Zeder C, Teles MJ, Porto G, Habermann JH, Dubach IL, Vallelian F, Frey BM, Moretti D, Baumgartner J, Zimmermann MB. The effect of a natural polyphenol supplement on iron absorption in adults with hereditary hemochromatosis. Eur J Nutr. 2022 Sep;61(6):2967-2977. doi: 10.1007/s00394-022-02829-8. Epub 2022 Mar 23. PMID 35320401